CLINICAL TRIAL: NCT01368783
Title: Two Randomized, Open-labeled, Parallel Designed Multiple-dose Clinical Trials to Evaluate Pharmacokinetics of Ritonavir-unboosted and Ritonavir-boosted Atazanavir Used Alone or Co-administered With Tenofovir DF in Healthy Korean and Caucasian Male Volunteers
Brief Title: Two Clinical Trials to Evaluate Pharmacokinetics of Unboosted and Boosted Atazanavir Used Alone or Co-administered With Tenofovir DF in Healthy Korean and Caucasian Male Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2011-ATV
Record Dates: First submitted 2011-06-07; First posted 2011-06-08 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-05

CONDITIONS: Atazanavir
MeSH Terms: interventions — Atazanavir Sulfate; Tenofovir; Ritonavir

ARMS (4):
- atazanavir (Experimental): 400 mg/day for 2 days
  Interventions: Drug: atazanavir
- Atazanavir and Tenofovir (Experimental)
  Interventions: Drug: Atazanavir(ATZ) and Tenofovir(TDF)
- Atazanavir and Ritonavir (Experimental)
  Interventions: Drug: Atazanavir(ATZ) + Ritonavir
- Atazanavir + tenofovir + ritonavir (Experimental)
  Interventions: Drug: atazanavir(ATZ) + tenofovir(TDF) + ritonavir

INTERVENTIONS:
Drug: atazanavir — 400 mg/day for 2 days
  Arms: atazanavir
Drug: Atazanavir(ATZ) and Tenofovir(TDF) — ATZ 400 mg with TDF/day for 2 days
  Arms: Atazanavir and Tenofovir
Drug: Atazanavir(ATZ) + Ritonavir — ATZ 300 mg + Ritonavir 100 mg/day for 2 days
  Arms: Atazanavir and Ritonavir
Drug: atazanavir(ATZ) + tenofovir(TDF) + ritonavir — ATZ 300 mg + Ritonavir 100 mg with TDF/day for 2 days
  Arms: Atazanavir + tenofovir + ritonavir

SUMMARY:
Compared to those of Caucasians, the plasma levels of atazanavir (ATV) may be higher in Koreans with the same dosage regimen(s). If so, even unboosted ATV could be used with tenofovir DF (TDF) which lowers the concentration of ATV. The investigators plan to investigate the pharmacokinetic features of ATV with or without TDF in healthy Korean and Caucasian volunteers and compare the ethnic differences.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 20 to 55 years old, with a weight more than 50 kg and with appropriate body mass index (BMI) values within 19-28 kg/m2.
* Agreed voluntarily to participate to the study and comply with the study protocol with written permission.

Exclusion Criteria:

* Has history of liver, kidney, respiratory, musculoskeletal, endocrinologic, neuropsychiatric, hemato-oncologic, or cardiovascular problem(s).
* Has history of hypersensitivity or clinically significant adverse drug reaction(s) to the study drugs, same class of the study drugs, or other drugs including aspirin and antibiotics.
* Drinks excessive caffeinated beverages (caffeine >10 units/day), alcohol beverages (alcohol >21 units/week) or smokes excessively (>20 cigarettes/day) or has history of alcoholism.
* Has been excluded by the researchers due to abnormal findings in screening EKG and/or blood tests

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2011-06

PRIMARY OUTCOMES:
Pharmacokinetic analysis
  maximum concentration at steady status(Cmax,ss)

SECONDARY OUTCOMES:
Pharmacokinetic evaluation
  Area under the time-concentration curve, at steady status, at tau(τ) (AUCτ,ss)

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Songpa-gu, Seoul, South Korea